CLINICAL TRIAL: NCT02156154
Title: Effect of Intravenous Acetaminophen on Postoperative Opioid-related Complications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Associate Staff Anesthesiologist, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-241
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous 0.9% sodium chloride (Placebo Comparator): 0.9% sodium chloride infusion will be initiated before the surgical incision with 100 ml and repeated every 6 hours for the earlier of 48 postoperative hours of hospital discharge.
  Interventions: Drug: Intravenous Acetaminophen
- Intravenous Acetaminophen (Experimental): Acetaminophen infusion will be initiated before the surgical incision with 1 g and repeated every 6 hours for the earlier of 48 postoperative hours of hospital discharge.
  Interventions: Drug: Intravenous Acetaminophen

INTERVENTIONS:
Drug: Intravenous Acetaminophen

SUMMARY:
Some patients have respiratory depression (decreased breaths per minute) after surgery. Acetaminophen, an FDA approved pain medication, may prevent this problem. The purpose of this study is to determine if acetaminophen decreases respiratory depression after surgery. The investigators will also evaluate the cost effectiveness of acetaminophen.

Patients having elective major abdominal surgery are being asked to participate in this research study. If eligible, a patient will have their baseline tidal volume (amount of air moved into or out of the lungs) and vital capacity (how much air the lungs are capable of holding) measured using a spirometer (apparatus for measuring the volume of air inspired and expired by the lungs) measured before surgery. Three questionnaires will also need to be completed before surgery.

The patient will then be randomized, like flipping a coin, to receive either Acetaminophen or placebo (inactive substance) as an infusion throughout surgery and for the first two days thereafter. Neither the patient nor his or her physician will know if the patient is assigned to study drug or placebo. Regardless of study assignment, both groups will receive standard pain management medications and sedation.

After surgery, the patient's blood pressure, activity, posture, respiratory rate, the electrical activity of the heart, oxygen saturation, tidal volume, minute ventilation and respiratory rate will be continuously monitored and recorded for 48 hours using a wireless pulse-oximeter and a respiratory volume monitor.

48 hours after surgery the patient will be asked to complete a patient satisfaction questionnaire, which will allow the patient to rate the satisfaction with the treatment received for pain. The patient will also be asked to complete a questionnaire about recovery.

At discharge, the patient will be given two questionnaires about pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18-85 years old
* above 50 kg
* American Society of Anaesthesiologists Physical Status 1-3
* Scheduled for elective open or laparoscopic abdominal surgery, including colorectal, prostate, and hysterectomy surgeries
* Patients with anticipated hospitalization of two nights
* Expected to require parenteral opioids for at least 48 hours for postoperative pain
* Able to use IV Patient-Controlled Analgesia systems

Exclusion Criteria:

* Hepatic disease, e.g. twice the normal levels of liver enzymes
* Kidney disease, e.g. twice the normal level of serum creatinine
* Epidural analgesia or regional blocks (including Transverse abdominis plane block)
* Acetaminophen sensitivity or known allergy
* Female patients who are pregnant or breastfeeding
* Patients taking warfarin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2014-12; Primary Completion 2019-03 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Turan A, Essber H, Saasouh W, Hovsepyan K, Makarova N, Ayad S, Cohen B, Ruetzler K, Soliman LM, Maheshwari K, Yang D, Mascha EJ, Ali Sakr Esa W, Kessler H, Delaney CP, Sessler DI; FACTOR Study Group. Effect of Intravenous Acetaminophen on Postoperative Hypoxemia After Abdominal Surgery: The FACTOR Randomized Clinical Trial. JAMA. 2020 Jul 28;324(4):350-358. doi: 10.1001/jama.2020.10009. PMID 32721009

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous 0.9% Sodium Chloride: 0.9% sodium chloride infusion will be initiated before the surgical incision with 100 ml and repeated every 6 hours for the earlier of 48 postoperative hours of hospital discharge.
  Intravenous Acetaminophen
- Intravenous Acetaminophen: Acetaminophen infusion will be initiated before the surgical incision with 1 g and repeated every 6 hours for the earlier of 48 postoperative hours of hospital discharge.
  Intravenous Acetaminophen
Period: Overall Study
Arm/Group | Intravenous 0.9% Sodium Chloride | Intravenous Acetaminophen
Started | 291 | 289
Completed | 287 | 283
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous 0.9% Sodium Chloride | Intravenous Acetaminophen | Total
Number analyzed (Participants) | 287 | 283 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (15.1) | 50.3 (15.3) | 49.3 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 140 | 276
  Male | 151 | 143 | 294
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 265 | 261 | 526
  Black | 15 | 14 | 29
  Other | 6 | 7 | 13
  Missing | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 287 | 283 | 570
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (4.8) | 26.7 (4.7) | 26.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hypoxemia
Description: Hypoxemia is measured as minutes with hypoxemia (Spo2 <90%) per hour of successful Spo2 monitoring. Patients will have nearly continuous pulseoximeter monitoring and recording. Data from the monitor will be downloaded daily for 48 hours postoperatively.
Time Frame: the initial 48 hours of postoperative monitoring or for the duration of hospitalization, if shorter.
Population: Patients were analyzed according to their randomized group, excluding patients who did not receive study intervention. 28 patients (5%) did not have any data recorded due to unexpected technical issues.
Measure: Median (Inter-Quartile Range); unit: min/h
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 283 | 287
min/h | 0.7 [0.1 to 5.1] | 1.1 [0.1 to 6.6]
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; A total of 28 patients (5%) were missing monitoring data (14 patients in each group). Values for these patients were obtained using multivariable imputation with 5 imputation data sets. The imputation regression model included all of the baseline, intraoperative, surgical, and postanesthesia care unit variables and all of the secondary outcomes; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney) — significance criterion of P < .044; Median Difference (Final Values) = -0.04, 95% CI 2-sided [-0.18 to 0.11] — Difference = IV Acetaminophen - Placebo group

2. Secondary Outcome: Time-weighted Pain Score During Initial 48 Postoperative Hours
Description: Pain scores were calculated on a visual analog scale of 0 to 10, with 0 being no pain and 10 being the most pain imaginable; time weighted mean was calculated as the area under the curve of the pain score measurements divided by total measurement time. Pain was recorded at roughly 15-minute intervals in the postanesthesia care unit and at 4-hour intervals on surgical wards
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: Data on the outcome could not be collected for 7 patients in the IV acetaminophen group and 5 patients in the IV sodium chloride group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 276 | 282
score on a scale | 4.2 (1.8) | 4.4 (1.8)
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.07, t-test, 2 sided — Confidence intervals were adjusted for 8 comparisons using Bonferroni correction (.05/8 = .006), for a significance criterion of P < .006; Mean Difference (Final Values) = -0.28, 99.4% CI 2-sided [-0.71 to 0.15] — Confidence intervals were adjusted for 8 comparisons using Bonferroni correction (.05/8 = .006), for a significance criterion of P < .006

3. Secondary Outcome: Time Weighted Pain Score in Post Anesthesia Care Unit
Description: Pain scores were calculated on a visual analog scale of 0 to 10, with 0 being no pain and 10 being the most pain imaginable; time-weighted mean was calculated as the area under the curve of the pain score measurements divided by total measurement time.
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: Data on the outcome could not be collected for 2 patients in the IV acetaminophen group and 6 patients in the IV sodium chloride group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 281 | 281
score on a scale | 4.3 (1.7) | 4.4 (1.8)
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.46, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.11, 99.4% CI 2-sided [-0.51 to 0.29] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Fatigue Score on Morning of Postoperative Day 1
Description: Fatigue scores were calculated on a scale of 1 to 10, with 1 being no fatigue and 10 being the worst fatigue imaginable.
Time Frame: Postoperative day 1
Population: Data on the outcome could not be collected for 12 patients in the IV acetaminophen group and 15 patients in the IV sodium chloride group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 271 | 272
score on a scale | 5 (2.6) | 4.9 (2.7)
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.56, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.13, 99.4% CI 2-sided [-0.49 to 0.76] — Treatment effect data are reported as differences in means between the study groups, assessed using a 2-sample t test

5. Secondary Outcome: Lowest RASS Score During Initial 48 Postoperative Hours
Description: Sedation was estimated by the RASS score and recorded at 2-hour intervals by ward nurses per clinical routine during the initial 48 postoperative hours. The Richmond Agitation-Sedation Scale (RASS) is scored from -5 to +4, with -5 being unarousable, 0 being alert and calm, and +4 being combative.
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: Data on the outcome could not be collected for 91 patients in the IV acetaminophen group and 86 patients in the IV sodium chloride group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 192 | 201
score on a scale | -0.96 (0.75) | -0.89 (0.76)
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -0.08, 99.4% CI 2-sided [-0.29 to 0.13] — Treatment effect data are reported as differences in means between the study groups, assessed using a 2-sample t test

6. Secondary Outcome: Time Spent in Sitting or Upright Position
Description: Treatment effect data are reported as ratios of geometric means
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: Data on the outcome could not be collected for 31 patients in the IV acetaminophen group and 37 patients in the IV sodium chloride group.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 252 | 248
hours | 2.2 [0.8 to 4.1] | 2.2 [0.9 to 4.2]
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.65, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Ratios of geometric means = 0.94, 99.4% CI 2-sided [0.63 to 1.39] — Treatment effect data are reported as ratios of geometric means, assessed using a 2-sample t test after logarithmic transformation of outcomes

7. Secondary Outcome: Opioid Consumption - Intravenous Morphine Equivalents
Description: Total opioid consumption over the initial 48 postoperative hours was extracted from patients' medical records and converted to intravenous morphine equivalents
Time Frame: Initial 48 postoperative hours
Population: Data on the outcome could not be collected for 3 patients in the IV acetaminophen group and 7 patients in the IV sodium chloride group.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 280 | 280
mg | 50 [18 to 122] | 58 [24 to 151]
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.22, t-test, 2 sided; Ratios of geometric means = 0.86, 99.4% CI 2-sided [0.61 to 1.21] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: Patients were asked about postoperative nausea and vomiting in the postanesthesia care unit, at 4-hour intervals while awake through the remaining initial day of surgery, and on the first and second postoperative mornings.
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 280 | 280
Participants | 140 | 124
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.18, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.13, 99.4% CI 2-sided [0.88 to 1.45] — Risk ratio = Treatment/Placebo

9. Secondary Outcome: Incidence of Low Respiratory Function Event
Description: A low respiratory function event was defined as an episode of less than 40% of predicted minute ventilation for 2 minutes.
Time Frame: Initial 48 postoperative hours or duration of hospitalization (whichever comes first)
Population: Data on the outcome could not be collected for 95 patients in the IV acetaminophen group and 124 patients in the IV sodium chloride group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 188 | 163
Participants | 52 | 50
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.53, Chi-squared — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 0.90, 99.4% CI 2-sided [0.57 to 1.43] — RR = Treatment/Placebo

10. Secondary Outcome: Total Anesthetic Dose From Induction to Extubation
Description: Total anesthetic dose is measured in minimal alveolar concentration hours.
Time Frame: Induction to extubation (3 hours on average)
Population: Data on the outcome could not be collected for 1 patient in the IV acetaminophen group.
Measure: Median (Inter-Quartile Range); unit: minimal alveolar concentration hours
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
Number analyzed (Participants) | 282 | 287
minimal alveolar concentration hours | 2.9 [2.6 to 3] | 2.9 [2.7 to 3]
Statistical Analysis 1: Comparison: Intravenous Acetaminophen vs Intravenous 0.9% Sodium Chloride; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney) — Adjusted for 8 comparisons using Bonferroni correction (.05/8 = .006), for a significance criterion of P < .006; Median Difference (Final Values) = 0, 99.4% CI 2-sided [-0.39 to 0.36] — Treatment effect is reported as median difference, estimated using the Hodges-Lehmann estimator of location shift

ADVERSE EVENTS:
Time Frame: 90 days
Description: No adverse events were recorded.
Arm/Group | Intravenous Acetaminophen | Intravenous 0.9% Sodium Chloride
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/287
Serious Adverse Events (participants affected / at risk) | 0/283 | 0/287
Other Adverse Events (participants affected / at risk) | 0/283 | 0/287

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02156154/Prot_SAP_000.pdf